CLINICAL TRIAL: NCT05268835
Title: Comparative Efficacy of Different Oral Doses of Clindamycin in Preventing Post-operative Sequelae of Lower Third Molar Surgery - a Randomized, Triple-blind Study
Brief Title: Different Oral Doses of Clindamycin in Preventing Post-operative Sequelae of Lower Third Molar Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oral and Maxillofacial Surgery Clinic, Poland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2022-02-24; First posted 2022-03-07 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Impacted Third Molar Tooth; Impacted Molar
Keywords: impacted third molars; post operative pain; trismus; infection
MeSH Terms: conditions — Pain, Postoperative; Trismus; Infections | interventions — Clindamycin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Clindamycin 150mg (Active Comparator): Patients receiving 150mg of clindamycin (Dalacin C, Pfizer) after surgery every 8 hours
  Interventions: Drug: Dalacin C
- Clindamycin 300mg (Active Comparator): Patients receiving 300mg of clindamycin after surgery every 8 hours
  Interventions: Drug: Dalacin C
- Clindamycin 600mg (Active Comparator): Patients receiving 600mg of clindamycin after surgery every 12 hours
  Interventions: Drug: Dalacin C

INTERVENTIONS:
Drug: Dalacin C — The objective of the intervention is to determine the effect of antibiotic prophylaxis with three different doses of clindamycin on preventing infection and other complications after surgical extraction of impacted mandibular third molars

SUMMARY:
The objective of the study is to determine the effect of antibiotic prophylaxis with three different doses of clindamycin on preventing infection and other complications after surgical extraction of impacted mandibular third molars.

DETAILED DESCRIPTION:
The objective of the study is to determine the effect of antibiotic prophylaxis with three different doses of clindamycin on preventing infection and other complications after surgical extraction of impacted mandibular third molars.

A randomized, triple blind, controlled clinical trial is conducted, in Oral and Maxillofacial Surgery Clinic. Patients were randomly allocated to three groups: I - receiving 150mg of clindamycin after surgery every 8 hours, II - receiving 300mg of clindamycin after surgery every 8 hours and III - receiving 600mg of clindamycin after surgery every 12 hours. Each group continued the therapy for five days. The investigators anticipate the overall decrease in risk of infection and other postoperative complications, however whether the differences between the clindamycin concentrations, occurrence of postoperative sequelae and pain in the three groups are statistically significant, remains to be seen.

ELIGIBILITY:
Inclusion Criteria:

* Child-bearing potential or non-child-bearing potential female or male, non-smoker, ≥ 18 and ≤65 years of age at the time of signing the informed consent, weighing >50kg.
* Non-child-bearing potential female subject is defined as follows:

  1. Post-menopausal state: absence of menses for 12 months prior to drug administration or hysterectomy with bilateral oophorectomy at least 6 months prior to drug administration.
  2. Surgically sterile: hysterectomy, bilateral oophorectomy, or tubal ligation at least 6 months prior to drug administration.
* Capable of consent.
* Patient scheduled to undergo the removal of bony impacted mandibular molar under short-acting local anesthetic (e.g. mepivacaine, articaine or lidocaine) preoperatively
* Patient who has signed a written informed consent obtained prior to any study-related procedures
* Patient able to understand and comply with protocol requirements and instructions
* Female patient of childbearing potential must be willing to use a highly efficient birth control method during the study

Exclusion Criteria:

* Clinically significant illnesses within 4 weeks prior to the administration of the study medication.
* Clinically significant surgery within 4 weeks prior to the administration of the study medication.
* Any clinically significant abnormality found during the medical screening.
* Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.
* Abnormal laboratory tests judged clinically significant.
* Positive testing for hepatitis B, hepatitis C, or HIV at screening.
* Electrocardiographic abnormalities (clinically significant) or vital sign abnormalities (systolic blood pressure lower than 90 over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or heart rate less than 50 or over 100 bpm) at screening.
* BMI≥ 30.0kg/m2.
* History of significant alcohol abuse within six months prior to the screening visit or any indication of the regular use of more than fourteen units of alcohol per week or positive alcohol breath test at screening. History of drug abuse or use of illegal drugs. Alcohol abuse is defined as the consumption of more than 90ml of liquor or spirits or 530ml of beer per day, for consecutive days during the 6-months period. Drug abuse is defined as any recreational drug for 5 consecutive days during the 6-month period.
* Patient with any known hypersensitivity to clindamycin or other related drugs (e.g., lincomycin), paracetamol or ibuprofen; having developed hypersensitivity reactions, including symptoms of asthma, rhinitis, angioedema or urticaria.
* History of allergic reactions to heparin.
* Use of any drugs known to induce or inhibit hepatic drug metabolism (examples of inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, rifampin/rifabutin; examples of inhibitors: antidepressants, cimetidine, diltiazem, erythromycin, ketoconazole, monoamine oxidase inhibitors, neuroleptics, verapamil, quinidine) within 30 days prior to administration of the study medication.
* Patient with current or chronic history of liver disease, or known hepatic or biliary abnormalities
* Patient with a current or chronic history of severe renal impairment
* Patient with severe heart failure (New York Heart Association (NHYA) Class IV)
* Patient with history of gastrointestinal bleeding or perforation, related to previous antibiotics or NSAIDs therapy; gastrointestinal haemorrhage, cerebrovascular haemorrhage or of other evolving haemorrhage; an active, or history of recurrent peptic ulcer/haemorrhage (two or more distinct episodes of proven ulceration or bleeding)
* Patient with inflammation or ulcerative disease of the oral mucosa
* Patient with known systemic lupus erythematosus
* Patient who undergoes an extraction of contralateral molar in the same procedure or a bony-impacted molar
* Patient treated by antibiotics, analgesics or nonsteroidal anti-inflammatory drugs (NSAIDs) within the 3 days prior to the day of randomization (or within 5 times the elimination half-life whichever the longest)
* Patient who received other antibiotics or analgesic than short-acting preoperative or intraoperative local anesthetic agents within 12 hours before the start of the surgery or peri-operatively until randomization
* Women with positive results on a urine pregnancy test or breastfeeding women or women of childbearing potential without an effective contraception
* Patient having any current dental or medical condition that could prevent safe participation in this study
* Unwillingness or inability to follow the procedures outlined in the protocol
* Use of prescription medication within 14 days prior to administration of study medication or over-the-counter products (including natural food supplements, vitamins, garlic as supplement) within 7 days prior to administration of study medication, except for topical products without systemic absorption.
* Difficulty to swallow study medication.
* Use of any tobacco products in the 90 days preceding drug administration.
* Any food allergy, intolerance, restriction or special diet that could, in the opinion of the Investigator, contraindicate the subjects' participation in this study.
* A depot injection or an implant of any drug within 3 months prior to administration of study medication.
* Subjects with a clinically significant history of tuberculosis, epilepsy, asthma, diabetes, psychosis, or glaucoma will not be eligible for this study.
* Clinically significant history of diarrhea subsequent to administration of antibacterial agents or antibiotics.
* Additional exclusion criteria for females only:

  1. Breast-feeding subject.
  2. Positive urine pregnancy test at screening
  3. Female subjects of childbearing potential having unprotected sexual intercourse with any non-sterile male partner (i.e., male who has not been sterilized by vasectomy for at least 6 months) within 14 says prior to study drug administration. Acceptable methods of contraception:

     1. condom + spermicide,
     2. diaphragm + spermicide,
     3. intra-uterine contraceptive device (placed at least 4 weeks prior to study drug administration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Post-surgical infectious complications. | Baseline - 60 minutes after administration
  May occur with one or more of the following: pain, fever, swelling, trismus, dry socket.
Post-surgical infectious complications. | 24 hours after surgery
  May occur with one or more of the following: pain, fever, swelling, trismus, dry socket.
Post-surgical infectious complications. | 48 hours after surgery
  May occur with one or more of the following: pain, fever, swelling, trismus, dry socket.
Post-surgical infectious complications. | 7 days after surgery
  May occur with one or more of the following: pain, fever, swelling, trismus, dry socket.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Janas-Naze, DMD,PhD,Prof, Principal Investigator — OMFS Clinic
Locations (1):
- OMFS Clinic, Zgierz, Poland

IPD SHARING:
Plan to Share IPD: Yes
If the results are published, the data will be stored at repository with doi.
Supporting Information: Study Protocol, CSR
Time Frame: in a year
Access Criteria: If the results are published, the data will be stored at repository with doi.